CLINICAL TRIAL: NCT05126186
Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide for Rescuing Patients With Graft Failure: a Phase II Study
Brief Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide for Rescuing Patients With Graft Failure
Acronym: HaploRescue
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200129
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Hematologic Diseases; Graft Failure; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- haplo-SCT with PTCy (Experimental): haploidentical (haplo) related donor Stem Cell Transplantation (haplo-SCT) with administration of post-transplantation cyclophosphamide (PTCy, which targets alloreactive T cells generated early after an HLA-mismatched transplant, sparing regulatory T cells and leaving unaffected the non-dividing hematopoietic stem cells)
  Interventions: Other: haplo-SCT with PTCy

INTERVENTIONS:
Other: haplo-SCT with PTCy — Conditioning regimen Fludarabine (30mg/m2/day from day -6 to day -4), Cyclophosphamide (14.5 mg/kg/day at day -6 and day -5) except for patients who received a total dose of Cyclophosphamide >100mg/Kg during the first Bone Marrow Transplantation Total Body Irradiation (2 Gray on day -1).
  Source of stem cell source Peripheral blood stem cell Minimal target dose of 4.106 CD34+ cells/kg of recipient
  GvHD prophylaxis Cyclophosphamide 50 mg/Kg/day at D+3 and D+4 Ciclosporine from day+5 (residual 200 à 300ng/l) Mycophenolate mofetyl at 15mg/Kg x2/day from day+5
  Prevention of EBV reactivation Rituximab : 150mg/m2 intravenously at Day+5 post Haplo-SCT Each infusion of Rituximab will be preceded by administration of anti-pyretic and an antihistaminic.

SUMMARY:
Prognosis of patients with graft failure is dismal, and re-transplantation is the sole option for long-term survival. Currently, there is no consensus concerning therapeutic options in patients with primary or secondary (within the 60 days post-transplantation) graft failure and finding a new donor within an acceptable delay is challenging. Literature is poor on the subject while the overall survival of such patients is about 30% at 1 year. This situation thus represents today a very challenging unmet medical need.

Recently, haploidentical (haplo) related donor Stem Cell Transplantation (haplo-SCT) have improved dramatically outcomes using T-cell replete grafts with administration of post-transplantation cyclophosphamide (PTCy, which targets alloreactive T cells generated early after an HLA-mismatched transplant, sparing regulatory T cells and leaving unaffected the non-dividing hematopoietic stem cells) and standard post-transplant immune suppression with a calcineurin inhibitor (CNI) and mycophenolate mofetil. Our group re-transplanted a patient who experienced two consecutive graft failures and was successfully managed through a third haplo-SCT from her son using PTCy. We then retrospectively collected and analyzed data from 26 primary graft failure patients transplanted between 2011 and 2017 in 15 centers on behalf of French Society for Stem Cell Transplantation and Cell Therapy (SFGM-TC). The study population consisted mainly of patients with primary or secondary (within the 60 days post-transplantation) graft failure who underwent haplo-SCT and received PTCy as graft-versus-host-disease prophylaxis. The 1-year overall survival was about 60% suggesting that this approach might be a valid option in this particular poor clinical situation but now need validation through a phase II multicenter, national, prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 3 to 70 years
* All hematological diseases
* Suffering from primary or secondary (within the 60 days post-transplantation) graft failure after a 1st allo-SCT
* With usual criteria for allo-SCT:

  * ECOG ≤ 2
  * No severe and uncontrolled infection
  * Cardiac function compatible with high dose of cyclophosphamide
  * Adequate organ function: ASAT and ALAT ≤ 2.5N, total bilirubin ≤ 2N, creatinine clearance ≥30ml / min
* With identification of a haploidentical donor (brother, sister, parents, adult children or cousin)
* Absence of donor specific antibody (DSA) detected in the patient with a MFI ≥ 1500 (antibodies directed towards the distinct haplotype between donor and recipient)
* With health insurance coverage (bénéficiaire ou ayant droit).
* Understand informed consent or optimal treatment and follow-up.
* Contraception methods must be prescribed during all the duration of the research. Women and men of childbearing age must use contraceptive methods within 12 months and 6 months after the last dose of cyclophosphamide, respectively.
* Having signed a written informed consent (2 parents for patients aged less than 18)

Exclusion Criteria:

* Aged< 3 years old and >70 years old
* With uncontrolled infection
* With Seropositivity for HIV or HTLV-1 or active hepatitis B or C defined by a positive PCR HBV or HCV and associated hepatic cytolysis
* Yellow fever vaccine within 2 months before transplantation
* Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix)
* Uncontrolled coronary insufficiency, recent myocardial infarction <6 month, current manifestations of heart failure, uncontrolled cardiac rhythm disorders, ventricular ejection fraction <50%
* Heart failure according to NYHA (II or more)
* Preexisting acute hemorrhagic cystitis
* Renal failure with creatinine clearance < 30ml / min
* Urinary tract obstruction
* Pregnant (β-HCG positive) or breast-feeding
* Who have any debilitating medical or psychiatric illness, which preclude understanding the inform consent as well as optimal treatment and follow-up
* COVID vaccination or recent COVID disease <3 months
* Tutorship or curatorship
* Contraindications to treatments used during the research

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | at one year

SECONDARY OUTCOMES:
Graft failure incidence | at 3 months
Neutrophils engraftment | at day 100
  3 consecutive days with neutrophiles >0.5 G/L
Platelets engraftment | at day 100
  7 consecutive days with platelets >20 G/L
Absolute numbers of neutrophils | at 1 month
Absolute numbers of neutrophils | at 2 months
Absolute numbers of neutrophils | at 3 months
Absolute numbers of neutrophils | at 6 months
Absolute numbers of neutrophils | at 12 months
Absolute numbers of neutrophils | through study completion, an average of 6 months
Absolute number of platelets | at one month
Absolute number of platelets | at 2 months
Absolute number of platelets | at 3 months
Absolute number of platelets | at 6 months
Absolute number of platelets | at 12 months
Absolute number of platelets | through study completion, an average of 6 months
Incidence of use of growth factors for poor hematopoietic reconstitution | at 3 months
Acute GvHD incidence | at 3 months
Chronic GvHD incidence | at 24 months
Relapse incidence | at 12 months
Relapse incidence | at 24 months
Progression free survival | at 12 months
Progression free survival | at 24 months
Incidence of CMV infection | at 12 months
Incidence of EBV infection | at 12 months
Incidence of severe infections | at 3 months
  Severe infections are defined as CTAE grade of 3 or 4
Incidence of severe infections | at 6 months
  Severe infections are defined as CTAE grade of 3 or 4
Incidence of severe infections | at 12 months
  Severe infections are defined as CTAE grade of 3 or 4
Incidence of severe infections | at 24 months
  Severe infections are defined as CTAE grade of 3 or 4
Incidence of veino-occlusive disease (VOD) | at 3 months
Severity of veino-occlusive disease (VOD) | at 3 months
Non-relapse mortality | at 24 months
Incidence of cardiac toxicities | at 12 months
Overall survival | at 24 months
Interval between first allo-SCT and rescue haplo-SCT | at 60 days
Quality of life for adults | at 3 months
  Quality of life will be assessed for adults using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for adults | at 6 months
  Quality of life will be assessed for adults using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for adults | at 12 months
  Quality of life will be assessed for adults using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for adults | at 24 months
  Quality of life will be assessed for adults using "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" EORTC QLQ-C30-V3 questionnaire.The QLQ-C30 is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life for minors | at 3 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning
Quality of life for minors | at 6 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning
Quality of life for minors | at 12 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning
Quality of life for minors | at 24 months
  Quality of life will be assessed for minor using The Pediatric Quality of Life Inventory™ (PedsQL™) The 36-item PedsQL™ Family Impact Module is a parent-report instrument designed to assess the impact of pediatric chronic health conditions on parents and the family. It includes 6 subscales measuring parents' self-reported functioning. The scale has five Likert response options, 'never', 'almost never', 'sometimes', 'often' and 'almost always' (corresponding to scores of 100, 75, 50, 25 and 0). Higher scores indicate better functioning
Proportion of patients with a donor chimerism of 90% or more | at 1 month
Proportion of patients with a donor chimerism of 90% or more | at 3 months
Proportion of patients with a donor chimerism of 90% or more | at 6 months
Proportion of patients with a donor chimerism of 90% or more | at 12 months
Immune reconstitution | at 3 months post-transplantation
  Immune reconstitution will be defined by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 6 months post-transplantation
  Immune reconstitution will be defined by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 12 months post-transplantation
  Immune reconstitution will be defined by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 24 months post-transplantation
  Immune reconstitution will be defined by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Iron overload estimation | at 3 months
Iron overload estimation | at 6 months
Iron overload estimation | at 12 months
Iron overload estimation | at 24 months

IPD SHARING:
Plan to Share IPD: Undecided